CLINICAL TRIAL: NCT04233086
Title: A Retrospective Observational Analysis of a Cohort With Heart Failure With Preserved Ejection Fraction From a BNP Pathway Clinic
Brief Title: Retrospective Observational Analysis of a Cohort With Heart Failure With Preserved Ejection Fraction
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Collaborators: Manchester Metropolitan University (Other)
Responsible Party: Sponsor
Other Study IDs: 262060
Record Dates: First submitted 2020-01-07; First posted 2020-01-18 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Heart Failure With Preserved Ejection Fraction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients referred through the BNP pathway: Patients throughout 2016 referred through the BNP pathway at Queen Alexandra Hospital will retrospectively be assessed for Reddy et al (2018) H2FPEF score.
  Interventions: Other: No intervention, observational only

INTERVENTIONS:
Other: No intervention, observational only — No intervention, observational only

SUMMARY:
Heart failure with preserved ejection fraction (HFpEF) is a complex condition with various causes that is not yet fully understood. Most significantly there is no single method of diagnosing or treating the condition. Recently a novel non-invasive diagnostic criterion to predict the likelihood of HFpEF was proposed called H2FPEF. The main limitation of this study was the use of a single centre population from the Mayo clinic in Rochester, US. Another limitation is that the H2FPEF diagnostic criterion consists of common and often co-existing conditions which could as a result overestimate HFpEF probability. The aim of the investigators is to retrospectively test the H2FPEF criteria on the population at Queen Alexandra Hospital (QAH) in Portsmouth, which is of a lower socio-economic status and greater ethnic diversity. Implications of the proposed project if H2FPEF is proved to be generalizable to the study population is that it can be used within the Trust and rolled out to others. This would allow diagnosis to be made quicker and more cost effectively using echocardiography and without the need for invasive cardiac catheterisation. On the other hand if H2FPEF is found not to be applicable to the population then further research would be required to find the ideal diagnostic tool.

DETAILED DESCRIPTION:
HFpEF was previously characterised as 'diastolic dysfunction' but this terminology was changed as it was found that diastolic dysfunction was also seen in patients with 'systolic dysfunction'. Myocardial stiffness which leads to increased filling pressures is a common pathophysiologic attribute of HFpEF despite its multifactorial aetiology. Other common conditions associated with HFpEF include: atrial fibrillation (AF), chronotropic incompetence, pulmonary hypertension, right ventricular dysfunction and endothelial dysfunction; with common non-specific risk factors such as: age, gender, hypertension, obesity, diabetes, metabolic syndrome and renal failure. This complex heterogeneity of HFpEF which is not yet fully understood highlights the difficulty that clinicians have in being able to diagnose the condition.

Diagnosis of HFpEF is difficult and as of yet there is no test to confirm diagnosis, with current guidelines saying initial diagnosis should include the presence of typical signs and symptoms, an elevated B-type natriuretic peptide (BNP) (>35 pg/mL and/or N-Terminal pro-B-type Natriuretic Peptide [NT-proBNP] >125 pg/mL) and ejection fraction ≥50%. Echocardiography is the preferred method of assessing for HFpEF due to it being widely available, non-invasive, and able to provide immediate results. Recent studies comparing the use of echocardiography against 'gold standard' invasive cardiac catheterisation to assess cardiac filling pressures found echocardiography to be just as accurate and reliable. Implications of this research would be that patients could be assessed as outpatients by focus echocardiography rather than invasively in the cardiac catheterisation lab, which would improve patient experience, enhance patient outcomes and prove cost-effective for trusts.

In response a recently proposed non-invasive diagnostic criteria called H2FPEF which assesses patients based on body mass index (BMI), the number of hypertensive medications they take, presence of AF, pulmonary pressure, age and filling pressure. The advantage of the H2FPEF score is that it uses only non-invasive echocardiography data alongside routine clinical data making it easy to derive. However one key limitation of their study is the population they used was all from the Mayo clinic and so the generalisability of their results has not been tested for other populations, such as those of lower socioeconomic status like in Portsmouth. A further limitation is the parameters chosen to create H2FPEF are all relatively common morbidities and usually co-exist, making it likely that it will over diagnose HFpEF.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-95yrs inclusive
* Currently or previously attended a heart failure clinic with a cardiology consultant at QAH
* Had an echocardiogram, ECG, BNP blood biomarker test in addition to a routine clinical evaluation (including age, weight and number of hypertensive medications) during January 1st 2016 - December 31st 2016.

Exclusion Criteria:

* Known structural heart disease
* Significant heart valve disease (greater than mild stenosis, greater than moderate regurgitation)
* Pulmonary arterial hypertension
* Constrictive pericarditis
* Pre-existing cardiomyopathy
* Heart transplantation

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants will be patients who have attended heart failure clinics at QAH between 01/01/2016 - 31/12/2016. Eligibility will be met by the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-04-03 (Actual)

PRIMARY OUTCOMES:
To assess the predictive and diagnostic accuracy of H2FPEF at predicting HFpEF on our patient population | February - April 2020
  Predictive accuracy calculated with logistic regression and diagnostic accuracy with specificity and sensitivity calculations

SECONDARY OUTCOMES:
Follow-up of patient outcomes - Hospital admissions | February - April 2020
  To assess number of hospital admissions after one year for the study population.
Follow-up of patient outcomes - Change in treatment | February - April 2020
  To assess any changes in treatment after one year for the study population.

CONTACTS AND LOCATIONS:
Overall Officials: Kaushik Guha, Principal Investigator
Locations (1):
- Portsmouth University Hospital, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No participant data will be shared under the Data Protection Act. Only overall results of the statistical analyses will be shared.

REFERENCES:
- [Background] Borlaug BA, Paulus WJ. Heart failure with preserved ejection fraction: pathophysiology, diagnosis, and treatment. Eur Heart J. 2011 Mar;32(6):670-9. doi: 10.1093/eurheartj/ehq426. Epub 2010 Dec 7. PMID 21138935
- [Background] Telles F, Marwick TH. Imaging and Management of Heart Failure and Preserved Ejection Fraction. Curr Treat Options Cardiovasc Med. 2018 Sep 27;20(11):90. doi: 10.1007/s11936-018-0689-9. PMID 30259312
- [Background] Borlaug BA. The pathophysiology of heart failure with preserved ejection fraction. Nat Rev Cardiol. 2014 Sep;11(9):507-15. doi: 10.1038/nrcardio.2014.83. Epub 2014 Jun 24. PMID 24958077
- [Background] Ferrari R, Bohm M, Cleland JG, Paulus WJ, Pieske B, Rapezzi C, Tavazzi L. Heart failure with preserved ejection fraction: uncertainties and dilemmas. Eur J Heart Fail. 2015 Jul;17(7):665-71. doi: 10.1002/ejhf.304. Epub 2015 Jun 16. PMID 26079097
- [Background] Harper AR, Patel HC, Lyon AR. Heart failure with preserved ejection fraction. Clin Med (Lond). 2018 Apr 1;18(Suppl 2):s24-s29. doi: 10.7861/clinmedicine.18-2-s24. PMID 29700089
- [Background] Lekavich CL, Barksdale DJ, Neelon V, Wu JR. Heart failure preserved ejection fraction (HFpEF): an integrated and strategic review. Heart Fail Rev. 2015 Nov;20(6):643-53. doi: 10.1007/s10741-015-9506-7. PMID 26404098
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Result] Reddy YNV, Carter RE, Obokata M, Redfield MM, Borlaug BA. A Simple, Evidence-Based Approach to Help Guide Diagnosis of Heart Failure With Preserved Ejection Fraction. Circulation. 2018 Aug 28;138(9):861-870. doi: 10.1161/CIRCULATIONAHA.118.034646. PMID 29792299
- [Result] Andersen OS, Smiseth OA, Dokainish H, Abudiab MM, Schutt RC, Kumar A, Sato K, Harb S, Gude E, Remme EW, Andreassen AK, Ha JW, Xu J, Klein AL, Nagueh SF. Estimating Left Ventricular Filling Pressure by Echocardiography. J Am Coll Cardiol. 2017 Apr 18;69(15):1937-1948. doi: 10.1016/j.jacc.2017.01.058. PMID 28408024
- [Result] Lancellotti P, Galderisi M, Edvardsen T, Donal E, Goliasch G, Cardim N, Magne J, Laginha S, Hagendorff A, Haland TF, Aaberge L, Martinez C, Rapacciuolo A, Santoro C, Ilardi F, Postolache A, Dulgheru R, Mateescu AD, Beladan CC, Deleanu D, Marchetta S, Auffret V, Schwammenthal E, Habib G, Popescu BA. Echo-Doppler estimation of left ventricular filling pressure: results of the multicentre EACVI Euro-Filling study. Eur Heart J Cardiovasc Imaging. 2017 Sep 1;18(9):961-968. doi: 10.1093/ehjci/jex067. PMID 28444160

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-04): https://cdn.clinicaltrials.gov/large-docs/86/NCT04233086/Prot_SAP_000.pdf